CLINICAL TRIAL: NCT06173063
Title: Safety and Effectiveness of A Novel Enteral Feeding System: Prospective Study.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated after the enrollment of 19 participants due to difficulties in recruitment (an enrollment of 25 participants was originally planned). No safety concerns were raised and no adverse events occurred.
Sponsor: Rockfield Medical Devices (Industry)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLP001
Record Dates: First submitted 2023-11-23; First posted 2023-12-15 (Actual); Results first posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Enteral Feeding
Keywords: Enteral Feeding; Mobility; Quality of Life; Elastomeric
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Intervention Model Description: 25 adult subjects from a screening population of 200
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Mobility+ Arm (Experimental): Adult patients using Mobility+ novel enteral feeding system for nutritional intake.
  Interventions: Device: Mobility+ Enteral Feeding System

INTERVENTIONS:
Device: Mobility+ Enteral Feeding System — Enteral feeding using a continuous feeding, self-powered, discreet, silent enteral feeding system.
  Other Names: Mobility+; MOB

SUMMARY:
The goal of this interventional study is to obtain information on the safety and effectiveness of a novel enteral feeding system in adult users requiring at least a portion of their nutritional intake via enteral feeding. The main questions it aims to answer are:

* Can the device be used safely and effectively?
* Does use of the device impact on patient's quality of life?

Participants will use Mobility+ enteral feeding system as their enteral feeding method for the duration of the study and will record their experiences.

DETAILED DESCRIPTION:
The study will allow 25 participants to use the Mobility+ system for their feeding sessions over the course of 14 consecutive days, following an initial 7-day period where participants have time to trial and get used to the new system. Participants' homes are the setting for the 21-day study duration.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Gastrostomy (G) tube or Jejunostomy (J) tubes
* Participant must require enteral tube feeding every day, as determined at the time of study enrolment
* Participant must use commercially available enteral formula with standard enteral feeding system(s) (gravity bag, bolus, pump or combination(s)), for some or all of their tube feeds, for daytime or day and night-time feeding
* Participant must be EN dependent i.e., 500 ml minimum daily feed intake from EN
* Participants must be able to swap from current system to Mobility+ for a minimum of two daily feeds per day for duration of study (Study days 1 -14)
* Participant must be >= 18 to reflect the subset of the intended use population being evaluated
* Participant must be willing to participate in the study and provide consent).
* Participants must have been on an enteral feeding regime for a minimum of 10 weeks
* Participants clinical functional capacity is adequate as determined by operator clinical judgement, to enable them to participate fully in the study
* Participants are suitable candidates for using Mobility+ as determined by operator clinical judgement on participant enteral feeding needs (as per prescription) and alignment with Mobility+ Flow Rate Guide

Exclusion Criteria:

* Participants who do not use commercially available enteral formula for some or all their formula needs
* Participants unable/unwilling to provide consent
* Participants whose enteral feeding needs do not match the offering of the Mobility+, as determined by operator clinical judgement
* Participants who have inadequate clinical functional capacity, as determined by operator clinical judgement to participate fully in the study e.g. neuromuscular or neurodegenerative disorders, or developmental delay
* Participants with very limited mobility, as determined by operator clinical opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Mundi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Cohort: This was a prospective, single arm, single-center, non-randomized, first in human, post-market clinical study.
Period: Overall Study
Arm/Group | Patient Cohort
Started | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patient Cohort
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Year] | 63.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kilogram] | 69.0 (15.0)
Height [Mean (Standard Deviation); unit: Centimetres] | 171.5 (9.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square metre] | 23.3 (3.4)
EN formula consumed [Mean (Standard Deviation); unit: milliliters per day] | 1174 (353)
EN daily calories [Mean (Standard Deviation); unit: kcal per day] | 1907 (553)
Daily EN feeding sessions [Mean (Standard Deviation); unit: Feeding sessions per day] | 2.9 (1.1)
Total infusion time [Mean (Standard Deviation); unit: hours per day] | 3.0 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Volume of Enteral Feed Consumed Per Day
Description: Volume in mls of enteral feed consumed in total, and with Mobility+
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: milliliters per day
Arm/Group | Patient Cohort
Number analyzed (Participants) | 17
milliliters per day
  Volume in milliliters of enteral feed consumed (Mobility+) | 1050 (363)
  Volume in milliliters of enteral feed consumed (other EN systems) | 256 (294)

2. Secondary Outcome: Patient Perspective on Mobility Using Current Enteral Feeding System vs Mobility+
Description: Subjective scale (Likert) - Ease of performing activities during feeding rated as: Very easy (5), Easy (4), Neutral (3), Difficult (2), Very difficult (1).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patient Cohort
Number analyzed (Participants) | 17
Scores on a scale
  Moving from one room to another (Baseline) | 2.6 (1.2)
  Moving from one room to another (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.6 (0.5)
  Going up and down stairs (Baseline) | 2.1 (1.3)
  Going up and down stairs (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.6 (0.5)
  Short walk (e.g 1 block) (Baseline) | 2.3 (1.2)
  Short walk (e.g. 1 block) (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.5 (0.6)
  Long walk (e.g. several blocks) (Baseline) | 1.9 (1.1)
  Long walk (e.g. several blocks) (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.4 (0.7)
  Travelling in car/public transport (Baseline) | 2.4 (1.2)
  Travelling in car/public transport (End of Study post 14 d feeding w/ Mobility+ (Day 21) | 3.8 (1.1)
  Moderate intensity physical activities (Baseline) | 1.8 (1.1)
  Moderate intensity physical activities (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 3.8 (1.0)
  Other daily activities (high intensity physical activities) (Baseline) | 1.8 (1.1)
  Other daily high intensity physical activities(End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 3.7 (0.9)
  Ability to sleep (Baseline) | 2.9 (1.5)
  Ability to sleep (End of Study End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 3.8 (1.1)
  Socializing with friends/family (Baseline) | 3.2 (1.1)
  Socializing with friends/family (End of Study End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.3 (0.8)

3. Secondary Outcome: Patient Perspective on Ease of Use Using Current Enteral Feeding System and Mobility+
Description: Subjective scale (Likert) - Ease of use of current enteral feeding systems and Mobility+ were rated as: Strongly agree (5), Somewhat agree (4), Neutral (3), Somewhat disagree (2), Strongly disagree (1).
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Patient Corhort: This was a prospective, single arm, single-center, non-randomized, first in human, post-market clinical study.
Arm/Group | Patient Corhort
Number analyzed (Participants) | 17
Scores on a scale
  System is easy to use (Baseline) | 3.8 (0.8)
  System is easy to use (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 3.5 (1.5)
  System is easy to carry (Baseline) | 2.8 (1.4)
  System is easy to carry (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.2 (1.0)
  The noise level of system is acceptable (Baseline) | 4.2 (1.2)
  The noise level of system is acceptable (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 4.8 (0.5)
  System allows me to feed discreetly (Baseline) | 1.9 (1.2)
  System allows me to feed discreetly (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 3.6 (1.3)
  I am satisfied with the overall performance of the system (Baseline) | 3.5 (1.2)
  I'm satisfied with overall system performance (End of Study post 14 d feeding w/ Mobility+ (Day 21)) | 3.6 (1.5)

4. Secondary Outcome: Patient Perspective on Feeding Intolerance Symptoms Experienced Using Current Enteral Feeding System and Mobility+
Time Frame: 14 days
Population: This data was not collected for operational reasons as it was considered over burdensome to ask participants these questions due to time pressures during study execution and the extent of questions already posed.
Arm/Group | Patient Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Participant Perspective on Quality of Life
Description: Subjective scale (Likert) - Perspective on Quality of Life rated as: Excellent (5), Good (4), Neutral (3), Bad (2), Very bad (1)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patient Cohort
Number analyzed (Participants) | 17
Scores on a scale
  Quality of life (participant perspective) at baseline | 3.6 (0.9)
  Quality of life (participant perspective) at end of Study, post 14 d feeding w/ Mobility+ (Day 21) | 3.7 (0.8)

6. Secondary Outcome: Usability of Mobility+ (Volume)
Description: Estimate if participants consume similar average volume of feed/day during the study, compared to baseline
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: milliliters per day
Arm/Group | Patient Cohort
Number analyzed (Participants) | 17
milliliters per day
  Total enteral feed volume consumed per day at baseline | 1174 (353)
  Total enteral feed volume consumed per day at end of Study, post 14 d feeding w/ Mobility+ (Day 21)) | 1306 (318)
  Total enteral feed kcal consumed per day, at baseline | 1848 (604)
  Total enteral feed kcal consumed per day, at study end, post 14 d feeding w/ Mobility+ (Day 21)) | 2034 (527)

7. Secondary Outcome: Usability of Mobility+ (kcal)
Description: Estimate if participants consume similar average kcals of feed/day during the study, compared to baseline
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: kcal per day
Arm/Group | Patient Cohort
Number analyzed (Participants) | 17
kcal per day
  Total enteral feed kcal consumed per day, at baseline | 1848 (604)
  Total enteral feed kcal consumed per day, at study end, post 14 d feeding w/ Mobility+ (Day 21)) | 2034 (527)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study (21 days).
Arm/Group | Patient Cohort
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT06173063/Prot_002.pdf
  • Statistical Analysis Plan (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT06173063/SAP_003.pdf